CLINICAL TRIAL: NCT06556810
Title: Phase 1b Pilot Study to Evaluate Atibuclimab (IC14) for Treatment of Acute Decompensated Heart Failure
Brief Title: IC14 for Treatment of Acute Decompensated Heart Failure
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Implicit Bioscience (Industry)
Collaborators: University of Virginia (Other); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC14HF01
Record Dates: First submitted 2024-08-08; First posted 2024-08-16 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Acute Decompensated Heart Failure
Keywords: Acute Decompensated Heart Failure; Congestive Heart Failure; Left Heart Failure; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — atibuclimab

STUDY DESIGN:
Intervention Model Description: Hospitalized patients with acute decompensated heart failure will be treated with an intravenous dose of IC14 and evaluated for safety, pharmacokinetics/pharmacodynamics, and preliminary clinic response
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IC14 (atibuclimab) (Experimental): 20 mg/kg intravenously once at baseline
  Interventions: Drug: Atibuclimab (IC14)

INTERVENTIONS:
Drug: Atibuclimab (IC14) — Atibuclimab (IC14) is a monoclonal antibody against human cluster of differentiation (CD)14, a key signaling molecule of the innate immune system
  Other Names: anti-CD14 monoclonal antibody

SUMMARY:
The goal of this clinical trial is to learn if drug atibuclimab (IC14) works to treat adults hospitalized with acute decompensated heart failure (ADHF). It will also learn about the safety of IC14. The main questions it aims to answer are:

Is the drug IC14 safe in patients with ADHF? What are the IC14 drug levels in the bloodstream after treatment with IC14? What is the impact of IC14 treatment on markers of disease in the bloodstream? What is the impact of IC14 treatment on measures of heart failure? There is no placebo arm in this study.

Participants will:

Take drug IC14 once via an intravenous infusion After the infusion, be visited in the hospital or visit the clinic 5 times for checkups and tests Answer questions about their medical status via a phone call 3 months after the infusion

DETAILED DESCRIPTION:
The proposed investigation is a pilot study to evaluate the safety and exploratory efficacy of IC14 administered via IV infusion in patients with ADHF.

The primary objective of this study is to determine safety of intravenous IC14 in patients acute decompensated heart failure. Exploratory biomarkers, clinical outcomes, and pharmacokinetic/pharmacodynamic measurements will be used to design further study of clinical efficacy of IC14 in the treatment of ADHF.

To characterize safety of IC14 administered via IV infusion, the following assessments are to be performed: treatment-emergent adverse events (AEs), safety laboratory studies, serious adverse events (SAEs), and presence of anti-drug antibodies.

To evaluate the effect of IC14, biomarkers including high-sensitivity C-reactive protein (hsCRP), B-type natriuretic peptide (BNP), urine sodium, and estimated glomerular filtration rate (eGFR) are measured at baseline and repeatedly after IC14 treatment. CRP is an established prognostic marker in heart failure that reflects systemic interleukin-6 as well as interleukin-1 activities. Measuring CRP area-under-the-curve allows for integrating measurements across multiple time points to quantify the acute inflammatory response more accurately.

Preliminary clinical efficacy will be measured by evaluating heart failure and cardiac performance outcomes at Day 10, including Dyspnea Visual Analogue Scale, Congestion Score, Doppler echocardiogram, non-invasive hemodynamics, bioimpedance analysis, cardiopulmonary exercise test and Kansas City Cardiomyopathy Questionnaire.

Pharmacokinetics will determine the serum concentration of IC14 over time. Pharmacokinetic measurements will be correlated with pharmacodynamic markers of IC14 biologic effect, including monocyte CD14 receptor occupancy.

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study only if they meet all of the following criteria:

1. Primary diagnosis for hospitalization is decompensated heart failure established as the finding at admission of both conditions listed below:

   1. dyspnea or respiratory distress or tachypnea at rest or with minimal exertion; and
   2. evidence of elevated cardiac filling pressure or pulmonary congestion (at least one of the conditions must be met):

      * Pulmonary congestion/edema a physical exam OR chest x-ray;
      * plasma BNP levels ≥200 pg/ml or N-terminal-proBNP ≥600 pg/ml; or
      * invasive measurement of left ventricular end-diastolic pressure (LVEDP) >18 mmHg or of pulmonary artery occluding pressure (wedge pressure) >16 mmHg.
2. The patient has a prior documentation of impaired left ventricular systolic function (left ventricular ejection fraction <40%) at most recent assessment by any imaging modality (within 12 months).
3. The patient is symptomatic for moderate to severe dyspnea at time of enrollment as indicated by a score on the visual analog scale for dyspnea of 40 or more (in a scale of 1 to 100, where 0 is no shortness of breath and 100 is extremely short of breath) in the prior 12 hours.
4. The patient has recently received (past 24 hours) or is scheduled to received intravenous loop diuretics.
5. The patient is of age ≥21 years old, willing and able to provide written informed consent and to comply with the protocol (i.e., reporting of symptoms).
6. The patient has screening plasma C-reactive protein levels >3 mg/L (0.3 mg/dL).
7. Males and females of childbearing potential must use effective contraception.

Exclusion Criteria:

1. The primary diagnosis for admission is NOT decompensated heart failure, including diagnosis of acute coronary syndromes, hypertensive urgency/emergency, tachy- or brady-arrhythmias.
2. Concomitant clinically significant comorbidities that would interfere with the execution or interpretation of the study including but not limited to acute coronary syndromes; uncontrolled hypertension or orthostatic hypotension; tachy- or brady-arrhythmias; acute or chronic pulmonary disease; or neuromuscular disorders affecting respiration.
3. Recent (previous 3 months) or planned cardiac resynchronization therapy (CRT) or valve surgeries.
4. Previous or planned implantation of left ventricular assist devices or heart transplant.
5. Current or planned use of intravenous inotropes.
6. Recent (<14 days) use of immunosuppressive or anti-inflammatory drugs (including oral corticosteroids at a prednisone equivalent dose of ≥0.5 mg/kg/day but not including inhaled or low-dose oral corticosteroids, non-steroidal anti-inflammatory drugs or colchicine).
7. Chronic inflammatory disorder (i.e., rheumatoid arthritis, systemic lupus erythematosus).
8. Active infection (of any type), including chronic/recurrent infectious disease (including hepatitis B virus, hepatitis C virus, and HIV/AIDS) - but excluding HCV+ with undetectable plasma RNA.
9. Active malignancy - excluding carcinoma in situ [any location] or localized non-melanoma skin cancer.
10. Any comorbidity limiting survival or ability to complete the study, including end-stage heart failure.
11. Stage V kidney disease or on renal-replacement therapy or renal transplant recipient.
12. Neutropenia (<1,500/mm3 or <1,000/mm3 in Black/African-American patients).
13. Pregnancy.
14. Hypersensitivity to IC14 or previous adverse reaction to antibody-based treatments.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety of IC14 treatment | 0-28 days
  safety measured by treatment-emergent adverse events, including abnormal laboratory values
Anti-Drug Antibodies following IC14 treatment | 0-28 days
  anti-drug antibodies

SECONDARY OUTCOMES:
C-reactive protein, biomarker of inflammation | baseline, 24 hours, 72 hours or discharge, Day 10, Day 29
  area under the curve (0 [normal]; 1-10 mg/dL [moderate elevation]; > 10 mg/dL [marked elevation] per time)
B-type natriuretic peptide, biomarker of heart failure | baseline, 24 hours, 72 hours or discharge, Day 10, Day 29
  absolute value (<100 pg/mL [normal], >=100 pg/mL [heart failure])
Estimated glomerular filtration rate, biomarker of heart failure | baseline, 72 hours or discharge, Day 10, Day 29
  absolute value(>=90 ml/min/1.73 m2 [normal]; 60-89 [possible impairment]; 15-59 [impairment]; <15 [renal failure])
Urine sodium | baseline, 24 hours, 72 hours or discharge
  absolute value (40-220 milliequivalents/day)
Dyspnea Visual Analogue Scale | baseline, 24 hours, 72 hours, Day 10, Day 29, and 3 months (virtual).
  10-cm Visual Analogue Scale
Congestion Score | baseline, 24 hours, 72 hours, Day 10, and Day 29
  a composite score of one point for peripheral edema, jugular venous distension ≥10 cm, pulmonary rales, or S3 gallop (0 [good] to 4 [poor])
Loop diuretic requirement | during the first 72 hours of hospitalization
  total loop diuretic requirement (in furosemide equivalents) as calculated from concomitant medication listings
Doppler echocardiogram | baseline, Day 10
  Change from baseline in left ventricular ejection fraction (left ventricular ejection fraction (>52% male, >54% female [normal])
Echocardiogram | baseline, Day 10
  Change from baseline in left ventricular global longitudinal strain (normal 21%)
Non-invasive hemodynamic assessment | baseline, 24 hours, 72 hours, Day 1
  Measure of cardiac output
Bioimpedance analysis | baseline, 24 hours, 72 hours, Day 1
  Measure of extracellular fluid as a marker of heart failure
Cardiopulmonary exercise test | Day 10
  aerobic exercise capacity (peak oxygen consumption [VO2]; <30 mL/kg/min [sedentary])
Pharmacokinetic determination of half-life, maximum concentration and area-under-the-curve | baseline, 15 minutes, 6 hours, 24 hours, 72 hours, Day 10, Day 29
  serum IC14 level
Pharmacodynamics | Day 10, Day 29
  Duration of monocyte CD14 receptor occupancy >90%
Ex-vivo leukocyte release assay | Day 10
  Lipopolysaccharide-stimulated release of interleukin 6
Kansas City Cardiomyopathy Questionnaire | baseline to 3 months
  Questionnaire for the patient that reports on 23 aspects of how heart failure affects the patient's life (0[worst symptoms/limitations]-100[least symptoms/limitations and excellent quality of life])

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Abbate, MD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - University of Virginia, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No